CLINICAL TRIAL: NCT00833482
Title: Study to Assess the Pharmacokinetic Drug - Drug Interactions Between Atazanavir Plus Ritonavir Coadministered With Voriconazole in Healthy Subjects
Brief Title: Drug Interactions Between Voriconazole and Atazanavir Coadministered as Atazanavir/Ritonavir in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: AI424-383; 2009-009095-13 (EudraCT Number)
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Results first posted 2012-10-25 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-09

CONDITIONS: Human Immunodeficiency Virus Type 1 (HIV-1); HIV Infections
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Voriconazole; Atazanavir Sulfate; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Voriconazole, 200 mg BID (EM) (Active Comparator)
  Interventions: Drug: Voriconazole
- Atazanavir/Ritonavir, 300/100 QD (EM & PM) (Active Comparator)
  Interventions: Drug: Atazanavir; Drug: Ritonavir
- Atazanavir/Ritonavir, 300/100mgQD + Voriconazole, 200mgBID(EM) (Active Comparator)
  Interventions: Drug: Voriconazole; Drug: Atazanavir; Drug: Ritonavir
- Voriconazole, 50 mg BID (PM) (Active Comparator)
  Interventions: Drug: Voriconazole
- Atazanavir/ritonavir, 300/100mgQD+voriconazole, 50mgBID (PM) (Active Comparator)
  Interventions: Drug: Voriconazole; Drug: Atazanavir; Drug: Ritonavir

INTERVENTIONS:
Drug: Voriconazole — Treatment A: Participants with functional CYP2C19 alleles (EM) received oral tablets of voriconazole, 400 mg, twice daily (BID), on Day 1, then 200 mg BID on Days 2 and 3. Voriconazole dose was given at least 1 hour after a light meal. Treatment C: EM participants received atazanavir/ritonavir, 300/100 mg once daily (QD), plus voriconazole, 400 mg BID on Day 21 then 200 mg BID on Days 22-30. Atazanavir/ritonavir dose was administered in the morning within 5 minutes of completing a light meal, and 1 hour before voriconazole morning dose. Treatment E: PM participants received atazanavir/ritonavir, 300/100 mg QD plus voriconazole, 100 mg BID, on Day 21, then 50 mg BID on Days 22-30.
  Arms: Atazanavir/Ritonavir, 300/100mgQD + Voriconazole, 200mgBID(EM); Atazanavir/ritonavir, 300/100mgQD+voriconazole, 50mgBID (PM); Voriconazole, 200 mg BID (EM); Voriconazole, 50 mg BID (PM)
Drug: Atazanavir — Treatment B in EM participants: EM participants received atazanavir/ritonavir, 300/100 mg once daily (QD), on Days 11 through 20. Treatment B in participants who were poor metabolizers of CYP2C19 (PMs): PM participants received oral tablets of atazanavir/ritonavir, 300/100 mg QD, on Days 11 through 20. Treatment C: EM participants received atazanavir/ritonavir, 300/100 mg QD, plus voriconazole, 400 mg BID on Day 21 then 200 mg BID on Days 22-30. Treatment E: PM participants received atazanavir/ritonavir, 300/100 mg QD plus voriconazole, 100 mg BID, on Day 21, then 50 mg BID on Days 22-30.
  Other Names: Reyataz; BMS-232632
  Arms: Atazanavir/Ritonavir, 300/100 QD (EM & PM); Atazanavir/Ritonavir, 300/100mgQD + Voriconazole, 200mgBID(EM); Atazanavir/ritonavir, 300/100mgQD+voriconazole, 50mgBID (PM)
Drug: Ritonavir — Treatment B: EM participants received atazanavir/ritonavir, 300/100 mg once daily (QD), on Days 11 through 20. Atazanavir/ritonavir dose was administered in the morning within 5 minutes of completing a light meal.
  Treatment C: EM participants received atazanavir/ritonavir, 300/100 mg QD, plus voriconazole, 400 mg BID on Day 21 then 200 mg BID on Days 22-30. Atazanavir/ritonavir dose was administered in the morning within 5 minutes of completing a light meal, and 1 hour before voriconazole morning dose.Treatment E: PM participants received atazanavir/ritonavir, 300/100 mg QD plus voriconazole, 100 mg BID, on Day 21, then 50 mg BID on Days 22-30. Treatment B in PM participants: PM participants received atazanavir/ritonavir, 300/100 mg QD, on Days 11 through 20. Atazanavir/ritonavir dose was administered in the morning within 5 minutes of completing a light meal.
  Arms: Atazanavir/Ritonavir, 300/100 QD (EM & PM); Atazanavir/Ritonavir, 300/100mgQD + Voriconazole, 200mgBID(EM); Atazanavir/ritonavir, 300/100mgQD+voriconazole, 50mgBID (PM)

SUMMARY:
This study assesses the effects of voriconazole, 200 mg, administered twice daily (BID), on the steady-state pharmacokinetics of atazanavir administered as atazanavir/ritonavir, 300/100 mg once daily (QD), in healthy participants with functional CYP2C19 alleles. The study also reviews the effects of atazanavir/ritonavir, 300/100 mg QD, on the pharmacokinetics of voriconazole, 200 mg, BID in healthy participants with functional CYP2C19 alleles.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants as determined by no clinically significant deviation from normal
* Body Mass Index (BMI) of 18 to 32 kg/m^2, inclusive. BMI=weight(kg)/height (m)^2
* Women who are not of childbearing potential (WOCBP)(ie, who are postmenopausal or surgically sterile) and men, ages 18 to 45 years, inclusive

Exclusion Criteria:

* WOCBP
* Sexually active fertile men not using effective birth control if their partners are WOCBP
* Proven or suspected acute hepatitis (within 12 months prior to the 1st dose)
* Any significant acute or chronic medical illness
* Any gastrointestinal surgery that could impact on the absorption of study drug
* Smoking more than 5 cigarettes per day
* History of any hemolytic disorders (including drug-induced hemolysis)
* History of acute or chronic pancreatitis
* History of hypochlorhydria or achlorhydria
* Men and women weighing <40 kg
* Positive blood screen for hepatitis C antibody, hepatitis B surface antigen, or HIV-1 or HIV-2 antibody
* Patients with galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 185 (Actual)
Dates: Start 2009-09; Primary Completion 2010-07 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- West Coast Clinical Trials, Llc, Cypress, California, United States
- Local Institution, Nijmegen, Netherlands

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 185 participants were enrolled in the study, and 153 were not treated, because they no longer met study criteria, withdrew consent, or were alternate participants who were no longer needed. The remaining 32 participants received treatment.
Groups:
- Voriconazole, 200 BID (EM): Participants with functional CYP2C19 alleles (EM) received voriconazole, 400 mg, twice daily (BID) on Day 1, then 200 mg BID on Days 2 and 3. Voriconazole dose was given at least 1 hour after a meal.
- Atazanavir/Ritonavir, 300/100 QD (EM): EM participants received atazanavir/ritonavir, 300/100 mg once daily (QD), on Days 11 through 20. Atazanavir/ritonavir dose was administered in the morning within 5 minutes of completing a light meal.
- Atazanavir/Ritonavir, 300/100mgQD + Voriconazole, 200mgBID(EM): EM participants received atazanavir/ritonavir, 300/100 mg QD, plus voriconazole, 400 mg BID on Day 21 then 200 mg BID on Days 22-30. Atazanavir/ritonavir dose was administered in the morning within 5 minutes of completing a light meal, and 1 hour before voriconazole morning dose.
- Voriconazole, 50 mg BID (PM): Participants who were poor metabolizers of CYP2C19 (PM)received voriconazole, 100 mg BID, on Day 1 then 50 mg BID on Days 2 and 3. Voriconazole dose was given at least 1 hour after a meal.
- Atanazivir/Ritonavir, 300/100 QD + Voriconazole, 50 BID (PM): PM participants received atazanavir/ritonavir, 300/100 mg QD, plus voriconazole, 100 mg BID, on Day 21, then 50 mg BID on Days 22-30.
- Atazanavir/Ritonavir, 300/100 QD (PM): PM participants received atazanavir/ritonavir, 300/100 mg QD, on Days 11 through 20. Atazanavir/ritonavir dose was administered in the morning within 5 minutes of completing a light meal.
Period: Days 1-3
Arm/Group | Voriconazole, 200 BID (EM) | Atazanavir/Ritonavir, 300/100 QD (EM) | Atazanavir/Ritonavir, 300/100mgQD + Voriconazole, 200mgBID(EM) | Voriconazole, 50 mg BID (PM) | Atanazivir/Ritonavir, 300/100 QD + Voriconazole, 50 BID (PM) | Atazanavir/Ritonavir, 300/100 QD (PM)
Started | 24 (Participants who received treatment) | 0 (Participants who received treatment) | 0 | 8 | 0 | 0
Completed | 24 | 0 | 0 | 8 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Days 11-20
Arm/Group | Voriconazole, 200 BID (EM) | Atazanavir/Ritonavir, 300/100 QD (EM) | Atazanavir/Ritonavir, 300/100mgQD + Voriconazole, 200mgBID(EM) | Voriconazole, 50 mg BID (PM) | Atanazivir/Ritonavir, 300/100 QD + Voriconazole, 50 BID (PM) | Atazanavir/Ritonavir, 300/100 QD (PM)
Started | 0 | 24 (Participants who received treatment.) | 0 | 0 | 0 | 8 (Participants who received treatment.)
Completed | 0 | 21 | 0 | 0 | 0 | 8
Not Completed | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Period: Days 21-30
Arm/Group | Voriconazole, 200 BID (EM) | Atazanavir/Ritonavir, 300/100 QD (EM) | Atazanavir/Ritonavir, 300/100mgQD + Voriconazole, 200mgBID(EM) | Voriconazole, 50 mg BID (PM) | Atanazivir/Ritonavir, 300/100 QD + Voriconazole, 50 BID (PM) | Atazanavir/Ritonavir, 300/100 QD (PM)
Started | 0 | 0 | 21 | 0 | 8 | 0
Completed | 0 | 0 | 20 | 0 | 7 | 0
Not Completed | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Extensive Metabolizers (EM): Participants with functional CYP2C19 alleles (extensive metabolizers, or EM).
- Poor Metabolizers (PM): Participants without a functional CYP2C19 allele (poor metabolizers, or PM).
- Total: Total of all reporting groups
Arm/Group | Extensive Metabolizers (EM) | Poor Metabolizers (PM) | Total
Number analyzed (Participants) | 24 | 8 | 32
Age Continuous [Mean (Standard Deviation); unit: years] | 31 (10) | 30 (7) | 31 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 20 | 8 | 28
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 2 | 8 | 10
  Black or African American | 1 | 0 | 1
  White | 20 | 0 | 20
  Not reported | 0 | 0 | 0
  Other | 1 | 0 | 1
CYP2C19 Genotype of Participants [Number; unit: Participants] — Genotypes with functional alleles indicative of extensive metabolizers=17/17, 1/17, 2/17, 3/17, 1/1, 1/2, and 1/3. Genotypes indicative of poor metabolizers=2/2, 2/3, and 3/3.
  Participants
    1/1 | 11 | 0 | 11
    1/2 | 5 | 0 | 5
    1/17 | 6 | 0 | 6
    2/2 | 0 | 6 | 6
    2/3 | 0 | 1 | 1
    2/17 | 1 | 0 | 1
    17/17 | 1 | 0 | 1
    3/3 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) and Minimum Observed Plasma Concentration (Cmin) of Atazanavir, Administered as Atazanavir/Ritonavir With and Without Voriconazole, in Participants Who Are Extensive Metabolizers (EM)
Description: EM participants are those with functional CYP2C19 alleles.
Time Frame: Predose and at 1, 2, 3, 4, 5, 7, 9,13, and 24 hours postdose on Days 20 and 30 of a 30-day cycle
Population: All participants who were healthy, who had functional CYP2C19 alleles, who received any study drug, and who had concentration-time data available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Atazanavir/Ritonavir, 300/100 QD (EM): Treatment B: EM participants received atazanavir/ritonavir, 300/100 mg once daily (QD), on Days 11 through 20. Atazanavir/ritonavir dose was administered in the morning within 5 minutes of completing a light meal.
- Atazanavir/Ritonavir, 300/100mgQD + Voriconazole, 200mgBID(EM): Treatment C: EM participants received atazanavir/ritonavir, 300/100 mg QD, plus voriconazole, 400 mg BID on Day 21 then 200 mg BID on Days 22-30. Atazanavir/ritonavir dose was administered in the morning within 5 minutes of completing a light meal, and 1 hour before voriconazole morning dose.
Arm/Group | Atazanavir/Ritonavir, 300/100 QD (EM) | Atazanavir/Ritonavir, 300/100mgQD + Voriconazole, 200mgBID(EM)
Number analyzed (Participants) | 22 | 20
ng/mL
  Atazanavir Cmin | 674 (61) | 525 (50)
  Atazanavir Cmax | 4715 (27) | 4076 (23)

2. Primary Outcome: Time to Maximum Concentration (Tmax) of Atazanavir, Administered as Atazanavir/Ritonavir With and Without Voriconazole, in EM Participants
Description: EM=extensive metabolizers, or participants with functional CYP2C19 alleles.
Time Frame: Predose and at 1, 2, 3, 4, 5, 7, 9,13, and 24 hours postdose on Days 20 and 30 of a 30-day cycle
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Atazanavir/Ritonavir, 300/100 QD (EM) | Atazanavir/Ritonavir, 300/100mgQD + Voriconazole, 200mgBID(EM)
Number analyzed (Participants) | 22 | 20
Hours | 3.0 [2.0 to 4.0] | 2.07 [2.0 to 4.0]

3. Primary Outcome: Area Under the Plasma Concentration-time Curve in 1 Dosing Interval [AUC(TAU)] of Atazanavir Administered as Atazanavir/Ritonavir With and Without Voriconazole, in EM Participants
Description: EM=extensive metabolizers, or participants with functional CYP2C19 alleles.
Time Frame: Predose and at 1, 2, 3, 4, 5, 7, 9,13, and 24 hours postdose on Days 20 and 30 of a 30-day cycle
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Atazanavir/Ritonavir, 300/100 QD (EM): Treatment B: EMs received atazanavir/ritonavir, 300/100 mg once daily (QD), on Days 11 through 20. Atazanavir/ritonavir dose was administered in the morning within 5 minutes of completing a light meal.
Arm/Group | Atazanavir/Ritonavir, 300/100 QD (EM) | Atazanavir/Ritonavir, 300/100mgQD + Voriconazole, 200mgBID(EM)
Number analyzed (Participants) | 22 | 20
ng*h/mL | 44634 (35) | 38276 (28)

4. Secondary Outcome: Cmax and Cmin of Ritonavir, Administered As Atazanavir/Ritonavir With and Without Voriconazole, in EM Participants
Description: Cmax=maximum observed plasma concentration; Cmin=minimum observed plasma concentration; EM=extensive metabolizers, or participants with functional CYP2C19 alleles.
Time Frame: Predose and at 1, 2, 3, 4, 5, 7, 9,13, and 24 hours postdose on Days 20 and 30 of a 30-day cycle
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Atazanavir/Ritonavir, 300/100 QD (EM) | Atazanavir/Ritonavir, 300/100mgQD + Voriconazole, 200mgBID(EM)
Number analyzed (Participants) | 22 | 20
ng/mL
  Ritonavir Cmax | 1597 (40) | 1429 (38)
  Ritonavir Cmin | 37.1 (61) | 28.3 (69)

5. Secondary Outcome: Tmax of Ritonavir, Administered As Atazanavir/Ritonavir With and Without Voriconazole, in EM Participants
Description: Tmax=time to maximum concentration; EM=extensive metabolizers, or participants with functional CYP2C19 alleles.
Time Frame: Predose and at 1, 2, 3, 4, 5, 7, 9,13, and 24 hours postdose on Days 20 and 30 of a 30-day cycle
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Atazanavir/Ritonavir, 300/100 QD (EM) | Atazanavir/Ritonavir, 300/100mgQD + Voriconazole, 200mgBID(EM)
Number analyzed (Participants) | 22 | 20
Hours | 4.0 [1.5 to 5.0] | 4.0 [2.0 to 4.0]

6. Primary Outcome: Tmax of Voriconazole, Administered With and Without Atazanavir/Ritonavir, in EM Participants
Description: Tmax=time to maximum concentration; EM=extensive metabolizers, or participants with functional CYP2C19 alleles.
Time Frame: Predose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours postdoseDays 3 and 30 of a 30-day cycle
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Groups:
- Voriconazole, 200 BID (EM): Treatment A: Participants with functional CYP2C19 alleles (EM) received voriconazole, 400 mg, twice daily (BID) on Day 1, then 200 mg BID on Days 2 and 3. Voriconazole dose was given at least 1 hour after a meal.
Arm/Group | Voriconazole, 200 BID (EM) | Atazanavir/Ritonavir, 300/100mgQD + Voriconazole, 200mgBID(EM)
Number analyzed (Participants) | 24 | 20
Hours | 1.50 [0.5 to 3.0] | 1.25 [1.0 to 3.0]

7. Primary Outcome: Cmax and Cmin of Voriconazole, Administered With and Without Atazanavir/Ritonavir, in EM Participants
Description: as for outcome 4
Time Frame: Predose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours postdoseDays 3 and 30 of a 30-day cycle
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Voriconazole, 200 BID: Treatment A: Participants with functional CYP2C19 alleles (EM) received voriconazole, 400 mg, twice daily (BID) on Day 1, then 200 mg BID on Days 2 and 3. Voriconazole dose was given at least 1 hour after a meal.
- Atazanavir/Ritonavir, 300/100mg QD + Voriconazole, 200 mg BID: Treatment C: EM participants received atazanavir/ritonavir, 300/100 mg QD, plus voriconazole, 400 mg BID on Day 21 then 200 mg BID on Days 22-30. Atazanavir/ritonavir dose was administered in the morning within 5 minutes of completing a light meal, and 1 hour before voriconazole morning dose.
Arm/Group | Voriconazole, 200 BID | Atazanavir/Ritonavir, 300/100mg QD + Voriconazole, 200 mg BID
Number analyzed (Participants) | 24 | 20
ng/mL
  Voriconazole Cmax | 3416 (49) | 3014 (47)
  Voriconazole Cmin | 776 (92) | 439 (144)

8. Primary Outcome: AUC(TAU)of Voriconazole, Administered With and Without Atazanavir/Ritonavir, in EM Participants
Description: AUC(TAU)=area under the plasma concentration-time curve in 1 dosing interval; EM=extensive metabolizers, or participants with functional CYP2C19 alleles.
Time Frame: Predose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours postdoseDays 3 and 30 of a 30-day cycle
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Voriconazole, 200 BID (EM) | Atazanavir/Ritonavir, 300/100mgQD + Voriconazole, 200mgBID(EM)
Number analyzed (Participants) | 24 | 20
ng.h/mL | 20284 (65) | 12944 (89)

9. Secondary Outcome: AUC(TAU) of Ritonavir, Administered As Atazanavir/Ritonavir With and Without Voriconazole, in EM Participants
Description: as for outcome 8
Time Frame: Predose and at 1, 2, 3, 4, 5, 7, 9,13, and 24 hours postdose on Days 20 and 30 of a 30-day cycle
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Atazanavir/Ritonavir, 300/100 QD (EM) | Atazanavir/Ritonavir, 300/100mgQD + Voriconazole, 200mgBID(EM)
Number analyzed (Participants) | 22 | 20
ng.h/mL | 9572 (37) | 8280 (32)

10. Secondary Outcome: Number of Participants With Death as Outcome, Serious Adverse Events (SAEs), Adverse Events (AEs) Leading to Discontinuation, and Any AE
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization.
Time Frame: Days 1 to 31 (discharge), continuously
Population: All participants who received study drug.
Measure: Number; unit: Participants
Groups:
- Atazanavir/Ritonavir, 300/100 QD (EM): Treatment B in EM participants: EM participants received atazanavir/ritonavir, 300/100 mg once daily (QD), on Days 11 through 20. Atazanavir/ritonavir dose was administered in the morning within 5 minutes of completing a light meal.
- Voriconazole, 50 mg BID (PM): Treatment D: Participants who were poor metabolizers of CYP2C19 (PM) received voriconazole, 100 mg BID, on Day 1 then 50 mg BID on Days 2 and 3. Voriconazole dose was given at least 1 hour after a meal.
- Atanazivir/Ritonavir, 300/100 QD + Voriconazole, 50 BID (PM): Treatment E: PM participants received atazanavir/ritonavir, 300/100 mg QD plus voriconazole, 100 mg BID, on Day 21, then 50 mg BID on Days 22-30.
- Atazanavir/Ritonavir, 300/100 QD (PM): Treatment B in PM participants: PM participants received atazanavir/ritonavir, 300/100 mg QD, on Days 11 through 20. Atazanavir/ritonavir dose was administered in the morning within 5 minutes of completing a light meal.
Arm/Group | Voriconazole, 200 BID (EM) | Atazanavir/Ritonavir, 300/100 QD (EM) | Atazanavir/Ritonavir, 300/100mgQD + Voriconazole, 200mgBID(EM) | Voriconazole, 50 mg BID (PM) | Atanazivir/Ritonavir, 300/100 QD + Voriconazole, 50 BID (PM) | Atazanavir/Ritonavir, 300/100 QD (PM)
Number analyzed (Participants) | 24 | 24 | 21 | 8 | 8 | 8
Participants
  Deaths | 0 | 0 | 0 | 0 | 0 | 0
  SAEs | 0 | 0 | 0 | 0 | 0 | 0
  AEs leading to discontinuation | 0 | 2 | 1 | 0 | 0 | 0
  Any AE | 22 | 24 | 21 | 0 | 3 | 2

11. Secondary Outcome: Number of Participants With Marked Abnormalities in Serum Chemistry Test Results
Description: LLN=lower limit of normal; ULN=upper limit of normal; preRX=pretreatment. Safety criteria: AST and ALT: If >1.25*ULN, or if preRX>ULN, use >1.25*preRX. Total and direct bilirubin: If >1.1*ULN or if preRX>ULN, use >1.25*preRX. Creatinine: If >1.33*preRX. Serum glucose, fasting: If preRX<LLN, use <.8*preRX or >ULN; if preRX>ULN, use >2*preRX or <LLN. Creatinine kinase: If >1.5*ULN or preRX>ULN, use >1.5*or preRX. Lactose dehydrogenase: If >1.25*ULN or preRX>ULN, use >1.5*preRX.
Time Frame: Within 21 days of Day 1 and on Days 3, 10, 20, 26, and 31 (at discharge)
Population: All participants who received study drug.
Measure: Number; unit: Participants
Groups:
- Atazanavir/Ritonavir, 300/100 QD + Voriconazole, 50 BID (PM): Treatment E: PM participants received atazanavir/ritonavir, 300/100 mg QD plus voriconazole, 100 mg BID, on Day 21, then 50 mg BID on Days 22-30.
Arm/Group | Voriconazole, 200 BID (EM) | Atazanavir/Ritonavir, 300/100 QD (EM) | Atazanavir/Ritonavir, 300/100mgQD + Voriconazole, 200mgBID(EM) | Voriconazole, 50 mg BID (PM) | Atazanavir/Ritonavir, 300/100 QD + Voriconazole, 50 BID (PM) | Atazanavir/Ritonavir, 300/100 QD (PM)
Number analyzed (Participants) | 24 | 24 | 21 | 8 | 8 | 8
Participants
  Aspartate aminotransferase (AST) (U/L): High | 0 | 0 | 1 | 0 | 0 | 0
  Alanine aminotransferase (ALT) (U/L): High | 0 | 1 | 1 | 0 | 1 | 1
  Total bilirubin (mg/dL): High | 4 | 22 | 21 | 0 | 8 | 7
  Direct bilirubin (mg/dL): High | 0 | 0 | 0 | 0 | 2 | 2
  Creatinine (mg/dL): High | 0 | 0 | 0 | 0 | 0 | 1
  Serum glucose, fasting (mg/dL): Low | 1 | 0 | 0 | 0 | 0 | 0
  Creatine kinase (U/L): High | 0 | 1 | 3 | 0 | 0 | 0
  Lactase dehydrogenase (U/L): High | 1 | 1 | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Marked Abnormalities in Hematology Laboratory Test and Urinalysis Results
Description: LLN=lower limit of normal; ULN=upper limit of normal; preRX=pretreatment. Safety criteria: Neutrophils + bands: If <.85*LLN or >1.15*ULN or ULN or if preRX<LLN, use <0.85*preRX or >ULN; if preRX>ULN, use >1.15*preRX or <LLN. Lymphocytes, relative: If <0.85*LLN or >1.15*ULN, or if preRX <LLN, use <0.85*preRX or >ULN; if preRX >ULN, use >1.15*preRX or <LLN. Blood, urine: If >= 2+, or if preRX >=1+, use >=2*preRX. White blood cells, urine: If >=2+, or if preRX >=2+, use >=4+. Red blood cells, urine: If >=2+ or if preRX >=2+, use >=4+. Not all categories were evaluated for each arm.
Time Frame: Within 21 days of Day 1 and on Days 3, 10, 20, 26, and 31 (at discharge)
Population: All participants who received study drug.
Measure: Number; unit: Participants
Groups:
- Voriconazole, 50 mg BID (PM): Treatment D: Participants who were poor metabolizers of CYP2C19 (PM)received voriconazole, 100 mg BID, on Day 1 then 50 mg BID on Days 2 and 3. Voriconazole dose was given at least 1 hour after a meal.
Arm/Group | Voriconazole, 200 BID (EM) | Atazanavir/Ritonavir, 300/100 QD (EM) | Atazanavir/Ritonavir, 300/100mgQD + Voriconazole, 200mgBID(EM) | Voriconazole, 50 mg BID (PM) | Atanazivir/Ritonavir, 300/100 QD + Voriconazole, 50 BID (PM) | Atazanavir/Ritonavir, 300/100 QD (PM)
Number analyzed (Participants) | 24 | 24 | 21 | 8 | 8 | 8
Participants
  Neutrophils + bands(absolute)(*10^3 cells/uL): Low | 1 | 0 | 1 | 0 | 0 | 0
  Lymphocytes, relative (*10*3 cells/uL): Low | 1 | 1 | 1 | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  Lymphocytes, relative (*10*3 cells/uL): High | 5 | 1 | 1 | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  Blood, urine: High | 1 | 1 | 2 | 0 | 0 | 0
  White blood cells (WBC), urine: High | 1 | 0 | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  Red blood cells (RBC), urine: High | 1 | 0 | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated

13. Secondary Outcome: Number of Participants With Investigator-identified Abnormalities in Electrocardiogram Results Not Present Prior to Administration of Study Drug and Considered Not Relevant and Not AEs by Investigator
Description: volt=voltage; LVH=left ventricular hypertrophy
Time Frame: Within 21 days of Day 1 and on Days -1, 21, and 31 (at discharge)
Population: All participants who received study drug.
Measure: Number; unit: Participants
Groups:
- Atanazivir/Ritonavir, 300/100 QD + Voriconazole, 50 BID (PM): Treatment E: PM participants received atazanavir/ritonavir, 300/100 mg QD, plus voriconazole, 100 mg BID, on Day 21, then 50 mg BID on Days 22-30.
Arm/Group | Voriconazole, 200 BID (EM) | Atazanavir/Ritonavir, 300/100 QD (EM) | Atazanavir/Ritonavir, 300/100mgQD + Voriconazole, 200mgBID(EM) | Voriconazole, 50 mg BID (PM) | Atanazivir/Ritonavir, 300/100 QD + Voriconazole, 50 BID (PM) | Atazanavir/Ritonavir, 300/100 QD (PM)
Number analyzed (Participants) | 24 | 24 | 21 | 8 | 8 | 8
Participants
  Sinus bradycardia | 0 | 0 | 0 | 0 | 2 | 0
  ST elevation and fusion complexes | 0 | 0 | 0 | 0 | 1 | 0
  T-wave abnormality + minimum volt criteria for LVH | 0 | 0 | 0 | 0 | 1 | 0
  Nonspecific T-wave abnormality | 0 | 0 | 0 | 0 | 1 | 0

14. Secondary Outcome: Number of Participants With Abnormalities in Vital Signs
Time Frame: Within 21 days of Day 1 and on Days -1, 1, 3, 11, 21, and 31 (at discharge)
Population: All participants who received study drug.
Measure: Number; unit: Participants
Arm/Group | Voriconazole, 200 BID (EM) | Atazanavir/Ritonavir, 300/100 QD (EM) | Atazanavir/Ritonavir, 300/100mgQD + Voriconazole, 200mgBID(EM) | Voriconazole, 50 mg BID (PM) | Atanazivir/Ritonavir, 300/100 QD + Voriconazole, 50 BID (PM) | Atazanavir/Ritonavir, 300/100 QD (PM)
Number analyzed (Participants) | 24 | 24 | 21 | 8 | 8 | 8
Participants
  Diastolic blood pressure | 0 | 0 | 0 | 0 | 0 | 0
  Systolic blood pressure | 0 | 0 | 0 | 0 | 0 | 0
  Heart rate | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory rate | 0 | 0 | 0 | 0 | 0 | 0
  Temperature | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Days 1 through 30, continuously, of a 30-day cycle.
Groups:
- Atazanazvir/Ritonavir, 300/100 QD + Voriconazole, 50 BID (PM): PM participants received atazanavir/ritonavir, 300/100 mg QD, plus voriconazole, 100 mg BID, on Day 21, then 50 mg BID on Days 22-30.
Arm/Group | Voriconazole, 200 BID (EM) | Atazanavir/Ritonavir, 300/100 QD (EM) | Atazanavir/Ritonavir, 300/100 QD (PM) | Atazanavir/Ritonavir, 300/100mgQD + Voriconazole, 200mgBID(EM) | Voriconazole, 50 mg BID (PM) | Atazanazvir/Ritonavir, 300/100 QD + Voriconazole, 50 BID (PM)
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/8 | 0/21 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 22/24 | 24/24 | 2/8 | 17/21 | 0/8 | 3/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Voriconazole, 200 BID (EM) (N=24) | Atazanavir/Ritonavir, 300/100 QD (EM) (N=24) | Atazanavir/Ritonavir, 300/100 QD (PM) (N=8) | Atazanavir/Ritonavir, 300/100mgQD + Voriconazole, 200mgBID(EM) (N=21) | Voriconazole, 50 mg BID (PM) (N=8) | Atazanazvir/Ritonavir, 300/100 QD + Voriconazole, 50 BID (PM) (N=8)
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0
Ocular icterus (Eye disorders) | 0 | 8 | 0 | 0 | 0 | 0
Chromatopsia (Eye disorders) | 2 | 0 | 0 | 2 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 6 | 1 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 0 | 3 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 12 | 3 | 0 | 2 | 0 | 0
Photophobia (Eye disorders) | 10 | 0 | 0 | 4 | 0 | 0
Fatigue (General disorders) | 2 | 4 | 0 | 3 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 8 | 1 | 0 | 5 | 0 | 0
Visual impairment (Eye disorders) | 5 | 1 | 0 | 3 | 0 | 0
Dizziness (Nervous system disorders) | 6 | 1 | 0 | 3 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 15 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 8 | 0 | 0 | 0 | 0
Scleral discolouration (Eye disorders) | 0 | 5 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Photopsia (Eye disorders) | 4 | 0 | 0 | 6 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.